CLINICAL TRIAL: NCT00936130
Title: Effect of Bariatric Surgery and Weight Loss on Energy Metabolism and Insulin Sensitivity "BARIA"
Brief Title: Bariatric Surgery and Weight Loss on Energy Metabolism and Insulin Sensitivity
Acronym: BARIA
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Eric Ravussin, p, Pennington Biomedical Research Center
Other Study IDs: PBRC 29004; Grant Number 25404 (Other Grant/Funding Number: Ethicon)
Record Dates: First submitted 2009-07-01; First posted 2009-07-09 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Obesity; Protein-energy; Imbalance; Insulin Sensitivity; Gastrointestinal Complication
Keywords: Roux-en-Y gastric bypass surgery; Sleeve gastrectomy (SGx) surgery; Gastric banding (GBx) surgery; Low calorie diet program
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Caloric Restriction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood draw, urine, stool, fat and muscle biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lifestyle counseling: This group will be comprised of participants on a low calorie diet program.
  Interventions: Behavioral: Low Calorie Diet
- Weight Loss Surgery: This group will be comprised of participants having weight loss surgery: Roux-en-Y gastric bypass, gastric banding, or sleeve gastrectomy.
  Interventions: Procedure: Laparoscopic Roux-en-Y gastric bypass; Procedure: Laparoscopic gastric banding; Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y gastric bypass — Laparoscopic Roux-en-Y gastric bypass surgery
  Other Names: RYGB
  Groups: Weight Loss Surgery
Procedure: Laparoscopic gastric banding — Laparoscopic gastric banding surgery
  Other Names: GBa
  Groups: Weight Loss Surgery
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy surgery
  Other Names: SGx
  Groups: Weight Loss Surgery
Behavioral: Low Calorie Diet — Low Calorie Diet Program
  Other Names: LCD
  Groups: Lifestyle counseling

SUMMARY:
The purpose of the study is to determine the effect of three weight loss surgeries compared to a low calorie diet with regard to energy expenditure, body composition, insulin sensitivity, and the response of gastrointestinal peptides to a standard meal. Baseline assessments will be conducted in all four groups and changes will be compared six and fifty-two weeks post-operatively.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effect of three weight loss procedures compared to a low calorie diet. Three different obesity surgery methods; Roux-en-Y gastric bypass (RYGB), gastric banding (GBa), sleeve gastrectomy (SGx), and one low calorie diet program on metabolism, with regard to body fat, physical activity levels, hormone changes after eating a meal, and changes in taste preferences.

Participants having obesity surgery will receive laparoscopic (minimally invasive surgery performed by making several small incisions in the abdomen and inserting a camera called a laparoscope) an adjustable gastric band, a sleeve gastrectomy or roux en Y gastric bypass. In addition to the regular surgical procedures, the surgeons will remove laparoscopically about 10g (1 tablespoon) of fat from within the abdomen. This fat tissue will be processed and stored for future study (at completion of the study) of your metabolism pre-treatment. Participants will complete post-operative follow-up appointments with their surgeon as required.

Participants on the LCD program will experience weight loss by following a low calorie diet program (LCD). For this diet you will select all your own food choices and our dietitians will assist you to reach your daily calorie target. You will be asked to follow this balanced food diet for the remainder of the 12 month study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ages of 18-65 years
* Body mass index >40 kg/m2 (BMI is calculated from your height and weight)
* BMI >35 kg/m2 with obesity associated diseases that should improve with weight loss (diabetes, hypertension, and sleep apnea)
* Medically qualified for obesity surgery by Drs LeBlanc or Hausmann

Exclusion Criteria:

* Women who are pregnant or unwilling to avoid pregnancy for 2 years post-operatively.
* Diabetes diagnosed more than 5 years ago
* Have had diabetes for more than 5 years
* Have had surgery on your stomach or intestinal tract except to remove your appendix or gall bladder.
* Have an active disease in your stomach or intestinal tract including inflammatory bowel disease.
* Have thyroid disease that is not treated
* Have any of the following psychiatric conditions that have not been treated to the point of complete remission: binge eating disorder, bulimia, current physical abuse, current sexual abuse, current substance abuse or dependence, mania or psychosis.
* Have any of the following psychiatric conditions that have not been treated to the point of partial remission prior to your enrollment in this study: anxiety, depression, dysfunctional marriage/family, personality disorder or post-traumatic stress disorder.
* Have a failure of one of your major organ systems. For example, liver failure, kidney failure, severe blood vessel blockage, or are not mentally able to understand the study and give your consent.
* Have a heart pacemaker or defibrillator, or any type of non-removable, metal containing objects in your body, as well as those with tattoos containing metallic dyes.
* Can not drink milk or products containing milk.
* Taking medications that alter your weight or metabolic rate. For example, antipsychotic drugs, beta adrenergic drugs (beta blockers), as well as anorectic drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medically qualified for obesity surgery by Drs LeBlanc or Hausmann
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Daily Energy Metabolism and insulin sensitivity | Enrollment, Baseline, Week 6-8 and Week 48-56 post-surgery / LCD diet
  Compare daily energy expenditure (accelerometry); body composition (EchoMRI, CT, MRS); insulin sensitivity (2-step hyperinsulinemic euglycemic clamp). Response of insulin, glucose, and gastrointestinal hormones. Changes in the stool microflora.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedial Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Broskey NT, Obanda DN, Burton JH, Cefalu WT, Ravussin E. Skeletal muscle ceramides and daily fat oxidation in obesity and diabetes. Metabolism. 2018 May;82:118-123. doi: 10.1016/j.metabol.2017.12.012. Epub 2018 Jan 4. PMID 29307520
- [Derived] Tam CS, Redman LM, Greenway F, LeBlanc KA, Haussmann MG, Ravussin E. Energy Metabolic Adaptation and Cardiometabolic Improvements One Year After Gastric Bypass, Sleeve Gastrectomy, and Gastric Band. J Clin Endocrinol Metab. 2016 Oct;101(10):3755-3764. doi: 10.1210/jc.2016-1814. Epub 2016 Aug 4. PMID 27490919
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151